CLINICAL TRIAL: NCT01871909
Title: Validation of LBNP Model of Human Hemorrhage in Trauma Patients
Brief Title: Validation of Lower Body Negative Pressure (LBNP) Model of Human Hemorrhage in Trauma Patients
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 13-0286
Record Dates: First submitted 2013-05-28; First posted 2013-06-07 (Estimated); Last update posted 2019-10-08 (Actual); Status verified 2019-10

CONDITIONS: Physical Trauma
Keywords: Physical trauma
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Physical trauma: Patients with report of physical trauma within 24 hours of presentation to the hospital.

SUMMARY:
Lower body negative pressure (LBNP) is a laboratory model used to study hemorrhage in humans. The investigators hypothesize that the physiologic changes that occur with application of LBNP mimic those observed in bleeding and hemodynamically unstable trauma patients, and that LBNP is a truly valid model of human hemorrhage.

DETAILED DESCRIPTION:
Specific aims:

1. Compare physiologic waveform data obtained from bleeding and hemodynamically unstable trauma patients to existing data collected from LBNP subjects.
2. Determine the accuracy of LBNP in approximating the physiologic changes that occur in bleeding and hemodynamically unstable trauma patients.

ELIGIBILITY:
Inclusion Criteria:

* age: 31 days - 89 years
* patients cared for in the Emergency Department (ED), Operating Room (OR), or the Intensive Care Unit (ICU) at Denver Health Medical Center, Children's Hospital Colorado and San Antonio Military Medical Center
* Patients with report of physical trauma within 24 hours of presentation at the hospital.

Exclusion Criteria:

* pregnant patients
* incarcerated patients
* patients who object at any time to participating in the study

Ages: 31 Days to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Trauma patients
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2013-10; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Waveform data comparison | Up to 12 months
  Compare physiologic waveform data obtained from bleeding and hemodynamically unstable trauma patients to existing data collected from LBNP subjects.
Approximation accuracy | Up to 12 months
  Determine the accuracy of LBNP in approximating the physiologic changes that occur in bleeding and hemodynamically unstable trauma patients.

CONTACTS AND LOCATIONS:
Overall Officials: Steve Moulton, MD, Principal Investigator — Children's Hospital Colorado
Locations (3):
- United States (3):
  - Children's Hospital Colorado, Aurora, Colorado
  - Denver Health Medical Center, Denver, Colorado
  - San Antonio Military Medical Center, San Antonio, Texas